CLINICAL TRIAL: NCT02999880
Title: Clinical Performance of Direct Anterior Composite Restorations Using Innovative Esthetic Dual-Shade Versus Polychromatic Natural Layering Technique Randomized Clinical Trial
Brief Title: Layering Technique Selection for Ultimate Aesthetics in Anterior Composites
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Ahmed Elzayat, principle investigator, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2016-10-237
Record Dates: First submitted 2016-12-08; First posted 2016-12-21 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Poor Aesthetics of Existing Restoration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Polychromatic layering (Control): (Experimental): Using and mixing different composite shades, opalescents and intensives.
  Interventions: Procedure: Polychromatic layering
- Dual-shade layering (Intervention): (No Intervention): Only two composite resin material shades the opaque dentin composite and enamel shade composite.

INTERVENTIONS:
Procedure: Polychromatic layering — Only two composite resin material shades will be used (opaque dentine composite and enamel shade composite).
  Arms: Polychromatic layering (Control):

SUMMARY:
the importance of this study is to evaluate the clinical performance of direct anterior resin composite restoration constructed using innovative esthetic dual-shade technique and another restoration constructed using polychromatic natural layering technique with various finishing and polishing steps.

The benefit from carrying out this study is to help the practitioners to decide the most suitable, easy, perfect technique to provide an optimally aesthetic, long lasting with superior clinical performance direct anterior resin composite restoration.

DETAILED DESCRIPTION:
-Study setting: Study is to be conducted in the Conservative Dentistry Department - Cairo University.

* Interventions:

  1. Preoperative clinical assessment:

     (O.S) will diagnose and select patients according to inclusion and exclusion criteria. He will record all base line data with understanding of patients' chief complains and aesthetic needs after treatment. Moreover, he will provide guidance for patients to prepare for the study.
     1. (A.H) and (G.Z) will take standard preoperative digital photographs before intervention by modifying mobile camera with smile lite (made in Switzerland) and smile capture 2016 contain 10 adaptors to allow connection between smile lite and the smartphone then photos will be saved in a computer.
     2. (A.H) and (G.Z) will take color shade using both Vita shade guide and Vita-Easy shade compact.
     3. .(A.H) and (G.Z) will ask patient for his satisfaction will be taken by visual analogue scale (0-100mm), 0 score refer to not satisfied at all, while 100 score refer to totally satisfied.
     4. (G.Z) and (A.H) will carry out all these tests at baseline, immediately after, 6 and 12 months in post-operative follow-up visits.
  2. Pre-operative planning (O.S) will be responsible for randomization according to patient selection for the sealed envelope containing which half will receive the control and the other will receive the intervention (Split mouth technique). Control group will be performed using polychromatic composite layering technique .Intervention group will be performed using dual shade composite layering technique.
  3. Intraoperative procedure: (G.Z) will do the following procedures:
* Silicone matrix will be fabricated either directly in the patient mouth using lingual surface of the remaining tooth structure and the existing restorations as a guide ,or fabricated on a study cast after optimizing the shape and function of the teeth with a wax up.
* Teeth preparation: after complete removal of caries a 1.5mm 75° functional- esthetic enamel bevel will prepared using 8888 diamond bur ( Brasseler, Savannah, GA, USA) on the facial surface, the lingual bevel will be 45° functional bevel, then a coarse disc (sof-lex,3M ESPE) will be used to extend the facial bevel where needed interproximally and toward the gingival third of the facial surface.
* Cleaning the teeth surface with fluoride-free paste(Depurdent, Dr Wild AG) and water.
* Teflon tape will placed on the adjacent teeth to prevent there being etched.

Application of each material is done according to the manufacture instructions:

* Application of 32% phosphoric acid (Uni-Etch,Bisco,Schaumburg, IL,USA) to enamel and dentine for 15 seconds.
* The acid etchant will then rinsed for 30 seconds, excess water will be eliminated and dental adhesive ( Adper Single Bond 2, 3M ESPE))will be applied.
* The silicon matrix will be seated followed by application of the lingual layer of composite( Filtek Supreme Ultra Universal Restorative[3M ESPE]) to form the lingual shell and after light curing the first increment the silicone matrix and Teflon tape will be removed.

Dual-shade layering (Intervention):

Only two composite resin material shades will be used (opaque dentine composite and enamel shade composite).

Polychromatic layering (Control):

Using and mixing different composite shades, opalescents and intensives.

* Finishing and polishing: will be performed using all grates of sof-lex discs (sof-lex,3M ESPE) , fine and Extra fine diamond burs (Brasseler), finishing strips, medium and fine rubber polishing points( Jiffy Polishers, Ultradent).

  d) Postoperative procedure:
* Patient satisfaction: using Visual analogue scale (0-100mm), 0 score refer to not satisfied at all, while 100 score refer to totally satisfied.
* Digital photographs using digital camera
* Color shade using Vita Easy shade:
* Clinical evaluation using FDI criteria:

(A.H) and (G.Z) will record all result outcomes on the following duration: immediately after, 6 and 12 months in post-operative follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for participants:

  1. Patients with good general health.
  2. Patients who will agree to the consent and will commit to follow-up period.
  3. Fully erupted anterior teeth with defects.
  4. Active caries, fractures, or defective Restorations in 6 anterior teeth.
  5. At least one spot lesion for contra-lateral anterior teeth on each side in the same jaw

Exclusion Criteria:

* Exclusion criteria for participants:

  1. Patients with any systemic disease that may affect normal healing.
  2. Patient with bad oral hygiene.
  3. Tetracycline or florsis staining.
  4. Patients who could/would not participate in all times of follow-up.
  5. Untreated periodontal disease was not allowed.
  6. Patients participating in more than 1 dental study.
  7. Patient received fluoride varnish during orthodontic treatment.
  8. Fully erupted anterior teeth with no defects.
  9. Patients with tendency to do bleaching during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2017-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | Change in satisfaction from baseline, after6 months and 0ne year
  Scale 0-100 cm, 0 is unsatisfied at all, 100 satisfied totally.

SECONDARY OUTCOMES:
Color shade | change in shade from baseline, after six months and one year
  Numerical

OTHER OUTCOMES:
Clinical performance including anatomic form, marginal discoloration,surface roughness, marginal adaptation and recurrent caries. | change from baseline, after six months and one year
  Numerical

IPD SHARING:
Plan to Share IPD: No